CLINICAL TRIAL: NCT02147262
Title: Inflammatory Proteins,Gene Polymorphisms, and Transcriptome Profiles in Patients With Chronic Atrophic Acrodermatitis
Brief Title: Laboratory Characteristics in Chronic Atrophic Acrodermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other); Medical University of Vienna (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Franc Strle, M.D., PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACA-0613
Record Dates: First submitted 2013-06-24; First posted 2014-05-26 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Chronic Atrophic Acrodermatitis
Keywords: chronic atrophic acrodermatitis; Lyme borreliosis; molecular characteristics; outcome
MeSH Terms: conditions — Lyme Disease | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACA-doxy 14 days (Active Comparator): patients with chronic atrophic acrodermatitis treated with doxycycline for 14 days
  Interventions: Drug: doxycycline orally, 100 mg, bid, 14 days
- ACA-doxy 28 days (Active Comparator): patients with chronic atrophic acrodermatitis treated with doxycycline for 28 days
  Interventions: Drug: doxycycline orally, 100 mg, bid, 28 days

INTERVENTIONS:
Drug: doxycycline orally, 100 mg, bid, 14 days
  Arms: ACA-doxy 14 days
Drug: doxycycline orally, 100 mg, bid, 28 days
  Arms: ACA-doxy 28 days

SUMMARY:
The main objective of this study is to characterize the inflammatory proteins, gene polymorphisms, and transcriptome profiles in patients with chronic atrophic dermatitis to gain better insight into pathogenesis of chronic infection with Borrelia burgdorferi sensu lato.

ELIGIBILITY:
Inclusion Criteria:

* chronic atrophic dermatitis in patients >18 years

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
inflammatory proteins in patients with chronic atrophic dermatitis | up to 24 months
  The inflammatory immune profiles will be assessed using Luminex to measure the expression of cytokines and chemokines representative of innate and adaptive TH1, TH2, TH17, and B cell responses.

SECONDARY OUTCOMES:
clinical characteristics of patients with chronic atrophic dermatitis treated with doxycycline for 14 or 28 days | at enrollment, at 2, 6 12 and 24 months follow-up

OTHER OUTCOMES:
gene polymorphisms in patients with chronic atrophic dermatitis | at enrollment, at 6 months follow-up
  The expression of disease-relevant genomic variants will be assessed using ImmunoChip.
transcriptome profiles in patients with chronic atrophic dermatitis | at enrollment
  We will use RNA sequencing of individual immune cell subtypes from patients to determine their transcriptome.

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, PhD, Study Chair — UMC Ljubljana; Dasa Stupica, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia